CLINICAL TRIAL: NCT04793542
Title: Evaluating Whether Lower-limb Hot Water Immersion Therapy Can Improve Symptoms in Individuals Diagnosed With Depression, Anxiety, and Post-traumatic Stress Disorders
Brief Title: Hot Water Immersion Therapy for Mental Health
Acronym: WITHME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lakehead University (Other)
Collaborators: Northern Ontario School of Medicine (Other)
Responsible Party: Principal Investigator, Nicholas Ravanelli, Assistant Professor, Lakehead University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1468218
Record Dates: First submitted 2021-03-04; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Anxiety Disorders; Depression; Post-traumatic Stress Disorder; Heat; Water Immersion
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention)
- Lukewarm Water (Sham Comparator)
  Interventions: Procedure: lower-limb hot water immersion
- Hot Water (Active Comparator)
  Interventions: Procedure: lower-limb hot water immersion

INTERVENTIONS:
Procedure: lower-limb hot water immersion — For a minimum of 30 minutes, 3 times a week for 8 consecutive weeks, participants will submerge their lower-limbs into 30-32°C (lukewarm) or 39-40°C (hot) water which will be measured with a supplied waterproof thermometer.
  Arms: Hot Water; Lukewarm Water

SUMMARY:
In 2016, it was estimated that nearly 1 billion people worldwide were affected by a mental or addictive disorder, and were associated with considerable excess mortality. Acute heat therapy sessions (e.g. whole-body heating or foot immersions) have been shown to improve symptoms in individuals diagnosed with common mental health illness such as major depressive disorders and reduce anxiety.

This study will assess the impact of an at-home 8-week lower-limb immersion in hot water on symptom severity in patients diagnosed with major depressive disorder, generalized anxiety disorder, and PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Diagnosed with depression, anxiety, or post-traumatic stress disorder
* Internet access (e.g. via smartphone, computer)
* Currently engaging in mental health treatment

Exclusion Criteria:

* Free of any mental health disorder
* Not engaging in regular mental health treatment
* Diagnosed with other psychiatric disorders (e.g. schizophrenia, bipolar disorder, panic disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire - 9 Item | Change from baseline at 8 weeks
  Self-report measure of depression severity
Change in General Anxiety Disorder - 7 Item | Change from baseline at 8 weeks
  Self-report measure of anxiety severity
Change in Post-Traumatic Stress Disorder Checklist - 20 Item | Change from baseline at 8 weeks
  Self-report measure that assesses symptoms of PTSD

SECONDARY OUTCOMES:
Post-water immersion thermal sensation | throughout study completion, 8 weeks in duration
  7-point scale to assess one's thermal state, with -3 defined as "Cold" and 3 defined as "Hot"
Post-water immersion thermal comfort | throughout study completion, 8 weeks in duration
  6-point scale to assess one's thermal satisfaction, with 1 and 6 defined as "very comfortable" and "very uncomfortable", respectively.
Post-water immersion thermal preference | throughout study completion, 8 weeks in duration
  5-point scale assessing whether the water temperature would be changed by the participant, with 2 defining 'much cooler' and -2 defining 'much warmer'

CONTACTS AND LOCATIONS:
Locations (1):
- Lakehead University, Thunder Bay, Ontario, Canada